CLINICAL TRIAL: NCT02169934
Title: A Study to Investigate the Metabolism and Excretion of [14C]-TRV130 Following Single Intravenous Dose Administration in Healthy Male Subjects
Brief Title: A Study to Investigate the Metabolism and Excretion of [14C]-TRV130 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP130-1007
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolabeled TRV130 (Experimental)
  Interventions: Drug: Radiolabeled TRV130

INTERVENTIONS:
Drug: Radiolabeled TRV130 — A single 2 mg IV dose administered as a 10 mL manual IV push over 2 minutes

SUMMARY:
The purpose of this study is to determine the routes of excretion for TRV130 and it's metabolites, and to determine and characterize, structurally, the metabolites present in plasma, urine, and feces in healthy male subjects.

DETAILED DESCRIPTION:
This study is an open-label, non-randomized, metabolism and excretion study of a single 2 mg IV dose of [14C] TRV130 (approximately 100 µCi) administered as a 10 mL manual IV push over 2 minutes in a fasted state.

ELIGIBILITY:
Key Inclusion Criteria:

* Males, between 18 and 64 years of age, inclusive
* With body weight ≥ 50 kg and body mass index (BMI) between 18 and 32 kg/m2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Negative test for selected drugs of abuse at Screening and at Check-in
* Able to comprehend and willing to sign an Informed Consent Form (ICF) prior to any study procedure
* A typical minimum of 1 to 2 bowel movements per day

Key Exclusion Criteria:

* History of sensitivity to any of the study medications or components thereof or a history of medication or other allergy that, in the opinion of the Investigator, contraindicates their participation
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 28 days prior to Check-in
* Participation in any other radiolabeled investigational study drug trial within 12 months prior to Check-in
* Exposure to significant radiation (eg, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to Check-in
* Has current malignancy, current systemic chemotherapy, or cancer diagnosis within 5 years prior to Screening (excluding squamous or basal cell carcinoma of the skin that has been clinically stable and fully excised in a curative procedure);
* Use of any tobacco- or nicotine-containing products within 6 months prior to Screening

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics (PK) of a single IV dose of [14C]-TRV130 | Day 1 - Day 13
To determine plasma concentrations of total radioactivity | Day 1 - Day 13
To determine whole blood concentrations of total radioactivity | Day 1 - Day 13
To determine urine concentrations of total radioactivity | Day 1 - Day 13
To determine fecal concentration of total radioactivity | Day 1 - Day 13

SECONDARY OUTCOMES:
To identify metabolites associated with TRV130 in blood, urine and feces | Day 1 - Day 13
Number of patients experiencing an Adverse Event | Day 1 - Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Trevena Inc, Study Director — Trevena Inc.
Locations (1):
- Madison Clinical Research Unit, Madison, Wisconsin, United States